CLINICAL TRIAL: NCT05422417
Title: New Form of Brain Stimulation Targeting Dorsomedial Prefrontal Cortex in Treating Refractory Depression and the Predictive Biomarkers of Antidepressant Efficacy
Brief Title: Dorsomedial Prefrontal Neuromodulation in Treatment-resistant Depression
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-TPEVGH No.: 2021-08-006A#1
Record Dates: First submitted 2022-06-07; First posted 2022-06-16 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Treatment-resistant Depression; Major Depressive Disorder
Keywords: rTMS; prolonged iTBS; brain stimulation; intermittent theta burst stimulation
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depressive Disorder, Major

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Prolonged intermittent theta-burst(iTBS)-DMPFC (Experimental): This active group will receive prolonged intermittent theta-burst(iTBS) on the dorsomedial prefrontal cortex(DMPFC)
  Interventions: Device: Prolonged intermittent theta burst stimulation (piTBS)
- 20Hz rTMS-DMPFC (Experimental): This active group will receive 20Hz rTMS on the DMPFC
  Interventions: Device: 20Hz rTMS
- Sham prolonged iTBS-DMPFC or 20Hz rTMS-DMPFC (Sham Comparator): Patients in the sham group will receive the same prolonged iTBS or 20Hz rTMS performed by a sham coil.
  Interventions: Device: sham control

INTERVENTIONS:
Device: Prolonged intermittent theta burst stimulation (piTBS) — Participants in the prolonged dosage (1800 pulse) of intermittent TBS (iTBS) active stimulation group will receive 2-week three-pulse 50-Hz bursts administered every 200 milliseconds (at 5 Hz) at an intensity of 80% active motor threshold (MT) to the bilateral DMPFC, twice a day. Stimulation will be delivered to the DMPFC using a stimulator.
  Arms: Prolonged intermittent theta-burst(iTBS)-DMPFC
Device: 20Hz rTMS — Participants in the 20 Hz rTMS (2000 pulse) active stimulation group will receive 2-week 2s- and-10s off, total 50 cycles at each hemisphere/session, at an intensity of 100% resting motor threshold (MT) to the bilateral DMPFC, twice a day. Stimulation will be delivered to the DMPFC using a stimulator.
  Arms: 20Hz rTMS-DMPFC
Device: sham control — Half of the patients in the sham group received 2-week the same prolonged iTBS parameter stimulation (sham- prolonged iTBS), and the other half received the same 20 Hz rTMS parameter stimulation using a sham coil (sham-20 Hz rTMS), which also improved the blinding process
  Arms: Sham prolonged iTBS-DMPFC or 20Hz rTMS-DMPFC

SUMMARY:
Major depressive disorder (MDD) is a common and troublesome disorder, with high risk of physical and psychiatric comorbidity. At least one-third of patients could not achieve a response after several antidepressant trials, so-called treatment-refractory depression (TRD). The high-frequency repetitive transcranial magnetic stimulation (rTMS) or intermittent theta-burst stimulation (iTBS) at left-sided dorsolateral prefrontal cortex (DLPFC) have a response rate of 40-60%. Obviously, not all TRD patients achieve the remitted state after treatment with antidepressants or DLPFC-rTMS, which may result from the heterogeneity of MDD. More and more evidence, such as brain lesion studies, deep brain stimulation, open-labeled rTMS case series, and neuroimaging studies, suggests that dorsomedial prefrontal cortex (DMPFC) might play a more central role in the pathophysiology of major depression. The DMPFC demonstrated as a "dorsal nexus" phenomenon in depression, which means a unique brain region where cortical networks for affect regulation, default mode control and cognitive control coverage in depressed subjects but not in healthy persons. In addition, another meta-analysis of resting-state functional MRI (fMRI) demonstrated the abnormal functional connectivity from DMPFC. These abnormalities of networks were highly associated with several depressive symptoms such as anhedonia, emotional regulation, somatic markers, rumination, self-reflection, poor attention and poor decision-making. However, only a handful of studies investigated the brain stimulation targeting DMPFC and the further changes in brain functional connectivity. The clinical efficacy and the fMRI changes of prolonged intermittent theta-burst stimulation (piTBS) and 20Hz- rTMS targeting bilateral DMPFC were investigated, and the predictive value of baseline networks by fMRI for antidepressant responses was also assessed to find a reliable approach to gauge treatment response prospectively.

DETAILED DESCRIPTION:
Several open label studies showed the preliminary clinical efficacy of DMPFC stimulation, but there was no randomized sham-control trial to confirm the clinical efficacy in Asian people. In addition, there were also few fMRI studies to express the brain circuit changes after DMPFC stimulation. The clinical efficacy and the fMRI changes of prolonged intermittent theta-burst stimulation (piTBS) and 20Hz- rTMS targeting bilateral DMPFC were investigated, and the predictive value of baseline networks by fMRI for antidepressant responses was also assessed to find a reliable approach to gauge treatment response prospectively. All patients with TRD who failed at least one antidepressant trial are randomized to three groups (Group-A: piTBS treatment; Group-B: 20Hz-rTMS treatment; Group-C: sham treatment). Before and after 20 sessions targeting bilateral DMPFC over ten days, structural and functional magnetic resonance imaging (MRI) is arranged for each participant. In addition, pre- and post-treatment fMRI data are analyzed for each patient to investigate the networks and local brain activity changes between groups.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a recurrent major depressive disorder based on Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV) criteria. Diagnoses were established after taking a thorough medical history and conducting a semistructured interview by administering the Mini International Neuropsychiatric Interview (MINI);
2. Recruited participants had to have a Clinical Global Impression - Severity score of at least four and a total score of at least 18 on the 17-items Hamilton Depression Rating Scale (HDRS-17);
3. Patients were qualified if they failed to respond to at least one adequate antidepressant treatment in their current episode (for example, failed to achieve 50% improvement of depression to an equivalent daily dose of 10 to 20 mg of escitalopram for at least eight weeks);
4. Stabilized treatment: keeping current antidepressant drug treatment, including the dose at least for four weeks before this trial and during the trial period; keep the stabilized psychotherapy at least for three months and no anticipated adjustment of types of psychotherapy and the frequency.

Exclusion Criteria:

1. Patients with Bipolar I and II disorder, schizophrenia, organic brain syndromes, or other major physical illnesses;
2. Patients who had received or will receive brain surgery or receive brain metal implantation (for example, neurostimulator) or received cardiac pacemakers;
3. Patients who had strong suicidal ideation within one week ( 3 points for third item of HDRS-suicidality)
4. Patients who had abnormal finding in the brain ( for example, brain tumor or arteriovenous malformation) or neurological disease ( for example, history of meningitis, encephalitis, epilepsy, stroke or neurodegenerative disease)
5. Pregnancy;
6. Patients who have metal implantation in the body, including cochlear implant, prosthetic heart valve, neurostimulator, clips.. etc
7. Patients who also failed to respond after receiving one completed course of electroconvulsive therapy (ECT) treatment or left dorsolateral prefrontal brain stimulation (adequate dose and adequate duration of ECT or DLPFC-rTMS and had followed up to monitor the efficacy at least for three months)
8. Claustrophobia for MRI screening;
9. Those who cannot follow the protocols, and did not sign informed consent proved by the institutional review board (IRB)

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2022-06-07 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in 17-item Hamilton Depression Rating Scale | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  the altered 17-item Hamilton Depression Rating Scale (range, 0 to 52, with higher scores indicating more depression)
Change in anxiosomatic cluster symptoms derived 17-item Hamilton Depression Rating Scale | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  the altered anxiosomatic cluster symptoms (range, 0 to 26, with higher scores indicating more severe anxiosomatic symptoms).The anxiosomatic cluster symptoms comprised nine items derived from HDRS-17: early insomnia, middle insomnia, slowness or retardation, psychic anxiety, autonomic anxiety, gastrointestinal symptoms, somatic symptoms, genital symptoms, and hypochondriasis.

SECONDARY OUTCOMES:
Response rate after 2-week treatment at the end of the trial, one month and three months after. | Time Frame: Week 2, Week 6(one month after brain stimulation), Week 14(three-month after brain stimulation)
  Improvement ≥ 50 % of 17-item Hamilton Depression Rating Scale (range, 0 to 52, with higher scores indicating more depression)
Remission rate after 2-week treatment at the end of the trial, one month and three months after. | Time Frame: Week 2, Week 6(one month after brain stimulation), Week 14(three-month after brain stimulation)
  17-item Hamilton Depression Rating Scale ≤7 (range, 0 to 52, with higher scores indicating more depression)
Changes in Clinical Global Index | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  Clinical Global Index, range from 1 to 7 with higher scores indicating worse clinical severity of illness.
Changes in depression severity, rated by self-reported | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  including Depression and Somatic Symptoms sub-scales, range from 0 to 66 with higher scores indicating more depressive and somatic symptom.
Changes in Young Mania Rating Scale | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  Young Mania Rating Scale, range from 0 to 60 with higher scores indicating more severe manic symptoms.
Baseline treatment refractory level and the further antidepressant efficacy of brain stimulation | Baseline and Week 2
  Maudsley staging method(MSM),, range from 3 to 15 with higher scores indicating higher treatment resistance.
Baseline treatment refractory level(TRDSS) and the further antidepressant efficacy of brain stimulation | Baseline and Week 2
  Treatment-resistant depression severity scale(TRDSS), range from 3 to 20 with higher scores indicating higher treatment resistance.
Baseline Life event stress scale and the further clinical efficacy of brain stimulation | Baseline and Week 2
  Life event stress scale,range from 0 to 1467 with higher scores indicating more life event stress.
Changes in depression severity, rated by Montgomery-Asberg Depression Rating Scale (MADRS) | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  the altered MADRS (range, 0 to 60 , with higher scores representing greater severity of depressive symptoms.
Change in Hamilton Anxiety Scale (HAMA) | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  the altered Hamilton Anxiety Scale (HAMA) (range, 0 to 56, with higher scores indicating more anxiety)
Baseline Rumination response scale (RRS) and the further clinical efficacy of brain stimulation | Baseline and Week 2
  RRS,range from 22 to 88 with higher scores indicating more rumination.
Change in Rumination response scale (RRS) | Time Frame: Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  RRS,range from 22 to 88 with higher scores indicating more rumination.
Baseline Snaith-Hamilton Pleasure Scale and the further clinical efficacy of brain stimulation | Baseline and Week 2
  The 14-item Snaith-Hamilton Pleasure Scale is a self-administered instrument. Each of the items has a set of four response categories--Definitely Agree, Agree, Disagree, and Strongly Disagree, with either of the Disagree responses receiving a score of 1 and either of the Agree responses receiving a score of 0. Thus, the SHAPS was scored as the sum of the 14 items so that total scores ranged from 0 to 14. A higher total SHAPS score indicated higher levels of present state of anhedonia.
Change in Snaith-Hamilton Pleasure Scale | Baseline, Week 1, Week 2, Week 3 (one week after brain stimulation), Week 6, Week 14(three-month after brain stimulation)
  The 14-item Snaith-Hamilton Pleasure Scale is a self-administered instrument. Each of the items has a set of four response categories--Definitely Agree, Agree, Disagree, and Strongly Disagree, with either of the Disagree responses receiving a score of 1 and either of the Agree responses receiving a score of 0. Thus, the SHAPS was scored as the sum of the 14 items so that total scores ranged from 0 to 14. A higher total SHAPS score indicated higher levels of present state of anhedonia.
Changes in EEG band before and after brain stimulation | Baseline and Week 2
  The value changes of prefrontal alpha, beta, theta, delta wave before and after 2 weeks treatment
Changes in brain connectivity before and after brain stimulation | Baseline and Week 2
  the change in resting-state functional connectivity
Changes in TMS-EEG/paired-pulse stimulation before and after brain stimulation | Baseline and Week 2
  the change in TMS-EEG/paired-pulse stimulation
Changes in cognitive performance of Taiwan Cognition Questionnaire | Baseline and Week 2
  Evaluate by Taiwan Cognition Questionnaire, range from 0 to 15 with higher scores indicating higher cognitive impairment
Changes in cognitive performance of word list recall. | Baseline and Week 2
  Evaluate by word list recall.
Changes in cognitive performance of Trail-Making Test | Baseline and Week 2
  Evaluate by Trail-Making Test
Changes in cognitive performance of Go/No-Go task | Baseline and Week 2
  Evaluate by Go/No-Go task
Changes in cognitive performance of Wisconsin Card Sorting Test | Baseline and Week 2
  Evaluate by Wisconsin Card Sorting Test

CONTACTS AND LOCATIONS:
Overall Officials: Chih-Ming Cheng, M.D., Principal Investigator — Taipei Veterans General Hospital, Taiwan
Locations (1):
- Taipei Veterans General Hospital, Taiwan, Taipei, Taiwan